CLINICAL TRIAL: NCT04738214
Title: Development of a Genome-based Platform for Personalized Treatment in Locally Advanced Rectal Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2020-1342
Record Dates: First submitted 2021-01-29; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: Rectal cancer, Personalized treatment, Genome-based platform, preoperative chemoradiotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Neoadjuvant CCRT+operation +/- adjuvant treatment — Patients receive neoadjuvant CCRT and operation. Adjuvant treatment after operation is performed depending on pathologic response. The patients showing pathologic complete response after neoadjuvant CCRT are not treated with any adjuvant treatment.

SUMMARY:
This study is aimed to develop a genome-based platform to predict patients who can achieve pathologic complete response after neoadjuvant treatment in locally advanced rectal cancer. The main treatments for locally advanced rectal cancer is surgical removal such as lower anterior resection after neoadjuvant CCRT. About 10-40% of patients showed pathologic complete response after neoadjuvant CCRT. Mandard tumor regression grade (TRG) is used to grade the histologic tumor response after neoadjuvant treatment. TRG 1 represents the pathologic complete response and TRG2 as histologically small group of cancer cells. Accordingly, TRG1 and 2 are expressed as good responder.

Even though the surgery is being performed as an essential treatment, there are various surgery-related sequelae such as colostomy. Also, in some patients, surgery may be refused or surgery may not be performed due to an underlying disease. About 15-20% of local recurrence was reported in patients who did not undergo surgery and the 3-year survival rate was 96.6%.

Colorectal cancer genetically can be divided into 4-subtypes. With the recent development of genome testing technology, genome analysis has been actively conducted in colorectal cancer. The most commonly known genetic subtype of colorectal cancer is classified into a total of 4 types as consensus molecular subtype (CMS); CMS1, CMS2, CMS3, CMS4. However, this was analyzed in colorectal cancer patients who did not undergo radiotherapy. There is no data regarding the response to radiation therapy according to each genetic subtype. Therefore, classifying the subtypes through genomic analysis and studying the responsiveness to radiotherapy in each subtype is needed.

In this study, we aimed to develop a platform that predicts pathologic tumor response after CCRT based on genomic information. Furthermore, being able to select patients who can wait-and-see without surgery using platform.

DETAILED DESCRIPTION:
The treatment in this study is one of the standard treatments suggested by the NCCN guidelines. The patients received operation after neoadjuvant concurrent chemoradiotherapy and pathologic tumor response is evaluated. Before neoadjuvant treatment, the following are obtained; Medical history and physical examination, Tissue acquisition through colonoscopy, Blood Test (CBC), Chemistry Test (SMA), staging through pelvic CT or MRI, PET-CT or chest CT.

Either 5-FU/leucovorin and Capecitabine based concurrent chemoradiotherapy is conducted. The target delineation is performed in 3mm simulation CT for radiotherapy. GTV includes primary lesions ,lymph nodes and mesorectum based on diagnostic CT, MRI, and PET-CT. CTV covers the perirectal and internal pelvic lymph node with microscopic margin of GTV. PTV1 is defined as extending 0.3cm from the GTV. PTV2 is defined as extending 0.5 from CTV. Radiotherapy is performed using 3D conformal radiotherapy, intensity-modulated radiotherapy, volumetric modulated Arc therapy. Radiotherapy is administered daily, five times a week according to the NCCN guidelines. Each treatment is performed with full bladder and prone positioning. Radiotherapy is performed 25 fractions with simultaneous integrated boost method. 2.00Gy is administered for PTV1 while 1.8 Gy is administered for PTV2.

The operation is performed 5-12 weeks after CCRT. If the patients refuse, physicians do not perform surgery and undergo wait-and-see. The treatment response is evaluated based on standard treatment process. During the treatment, the regular check up is conducted to evaluate the acute toxicity regarding treatment.

The acquired specimens are used for RNA sequencing and organoid construction. The RNA sequencing is used to analyze the differentially expressed based on treatment response to neoadjuvant concurrent chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 19 years old
2. Clinically or histologically diagnosed rectal cancer (adenocarcinoma)
3. Patients who satisfy all of the following conditions with either rectal cancer stage T3-4 or T2 in lower rectal cancer with any N stage according to 8th edition of American Joint Committee on Cancer

   - Stage T3-4 (T2 in lower rectum) in CT or MRI
4. Performance status 0 or 1 based on ECOG
5. Patients agreed to provide the tissue sample
6. Diseases can be evaluated according to RECIST Version 1.1
7. Patients who voluntarily agreed to informed consent

Exclusion Criteria:

1. Patients with distant metastasis
2. Patients with uncontrolled viral infection (HIV, HBV, HCV)
3. Patient who are pregnant, or have possibility of pregnancy and are on lactating
4. Hypersensitivity or history of allergic to the drug being used
5. Patients with cerebrovascular disease, complications, and infections that are not medically controlled
6. Patients with history of other malignant diseases within the past 5 years (excluding cured non-melanoma skin cancer or in situ cervical cancer)
7. Those who are taking drugs that can cause drug interactions with chemotherapy
8. Patients who withdraw consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced rectal cancer are subject to this trial. The patients undergo endoscopic biopsy and receive neoadjuvant CCRT and surgery. In case that pathologic CR status obtained after CCRT, no additional treatment is performed. Patients without pathologic CR status are treated with adjuvant treatment.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2025-01-18 (Estimated); Study Completion 2025-01-18 (Estimated)

PRIMARY OUTCOMES:
Pathologic response rate | up to 2 year
  The rate of patients who achieved complete response or partial response after concurrent chemoradiotherapy

SECONDARY OUTCOMES:
Disease free survival | up to 2 year
  The rate of patients without disease or death after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Woong Sub Koom, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Research related documents will be stored in a file with a separate password under the responsibility of the lead researcher and stored in a locked laboratory. These research-related records will be kept for 3 years from the time the research is completed, and after that, the research team will discard the documents.
  Tissue samples obtained from patients are subjected to genome analysis by extracting RNA and DNA. Patient registration information is encrypted and stored separately, and stored in freezer at -80°C until experimentation at Yonsei University Medical Research Institute under the supervision of the research director.

REFERENCES:
- [Background] Glynne-Jones R, Wyrwicz L, Tiret E, Brown G, Rodel C, Cervantes A, Arnold D; ESMO Guidelines Committee. Rectal cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2017 Jul 1;28(suppl_4):iv22-iv40. doi: 10.1093/annonc/mdx224. No abstract available. PMID 28881920
- [Background] Martens MH, Maas M, Heijnen LA, Lambregts DM, Leijtens JW, Stassen LP, Breukink SO, Hoff C, Belgers EJ, Melenhorst J, Jansen R, Buijsen J, Hoofwijk TG, Beets-Tan RG, Beets GL. Long-term Outcome of an Organ Preservation Program After Neoadjuvant Treatment for Rectal Cancer. J Natl Cancer Inst. 2016 Aug 10;108(12):djw171. doi: 10.1093/jnci/djw171. Print 2016 Dec. PMID 27509881
- [Background] Scott JG, Berglund A, Schell MJ, Mihaylov I, Fulp WJ, Yue B, Welsh E, Caudell JJ, Ahmed K, Strom TS, Mellon E, Venkat P, Johnstone P, Foekens J, Lee J, Moros E, Dalton WS, Eschrich SA, McLeod H, Harrison LB, Torres-Roca JF. A genome-based model for adjusting radiotherapy dose (GARD): a retrospective, cohort-based study. Lancet Oncol. 2017 Feb;18(2):202-211. doi: 10.1016/S1470-2045(16)30648-9. Epub 2016 Dec 18. PMID 27993569